CLINICAL TRIAL: NCT03330405
Title: A PHASE 1B/2 STUDY TO EVALUATE SAFETY AND ANTI TUMOR ACTIVITY OF AVELUMAB IN COMBINATION WITH THE POLY(ADENOSINE DIPHOSPHATE [ADP]-RIBOSE) POLYMERASE (PARP) INHIBITOR TALAZOPARIB IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: Javelin Parp Medley: Avelumab Plus Talazoparib In Locally Advanced Or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the investigational treatments have been moved to a continuation study (NCT05059522).
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B9991025; 2017-001509-33 (EudraCT Number); JAVELIN PARP MEDLEY (Other: Alias Study Number)
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Avelumab in Combination With Talazoparib Will be Investigated in Patients With Locally Advanced (Primary or Recurrent) or Metastatic Solid Tumors
Keywords: NSCLC, TNBC, hormone receptor positive (HR+) breast cancer, recurrent epithelial ovarian cancer, UC, and castration resistant prostate cancer (CRPC).
MeSH Terms: conditions — Recurrence; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Carcinoma, Ovarian Epithelial | interventions — avelumab; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Dose Level 0 Phase 1b (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 1b; Drug: Talazoparib Phase 1b
- Dose Level -1 Phase 1b (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 1b; Drug: Talazoparib Phase 1b
- Dose Level -2 Phase 1b (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 1b; Drug: Talazoparib Phase 1b
- A1. NSCLC Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- A2. NSCLC PD-L1 Resistant DDR+ Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- B1. TNBC Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- B2. HR+BC DDR Defect +Assay Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- C1. Ovarian CA Recurrent Plat-Sensitive Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- C2.Ovarian CA Recurrent Plat-Sensitive BRCA defect Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- D.Urothelial CA Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- E1. CRPC Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- E2. CRPC DDR Defect +Assay Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2
- F: Advanced Solid Tumors with BRCA or ATM defect Phase 2 (Experimental): Drug: Avelumab
  Drug: Talazoparib
  Interventions: Drug: Avelumab Phase 2; Drug: Talazoparib Phase 2

INTERVENTIONS:
Drug: Avelumab Phase 1b — Avelumab
  Other Names: MSB0010718C
  Arms: Dose Level -1 Phase 1b; Dose Level -2 Phase 1b; Dose Level 0 Phase 1b
Drug: Talazoparib Phase 1b — Talazoparib
  Other Names: MDV3800, BMN 673
  Arms: Dose Level -1 Phase 1b; Dose Level -2 Phase 1b; Dose Level 0 Phase 1b
Drug: Avelumab Phase 2 — The dose will be determined after the overall available data (including safety and preliminary anti tumor activity) emerging from the Phase 1b portion of the study have been evaluated.
  Other Names: MSB0010718C
  Arms: A1. NSCLC Phase 2; A2. NSCLC PD-L1 Resistant DDR+ Phase 2; B1. TNBC Phase 2; B2. HR+BC DDR Defect +Assay Phase 2; C1. Ovarian CA Recurrent Plat-Sensitive Phase 2; C2.Ovarian CA Recurrent Plat-Sensitive BRCA defect Phase 2; D.Urothelial CA Phase 2; E1. CRPC Phase 2; E2. CRPC DDR Defect +Assay Phase 2; F: Advanced Solid Tumors with BRCA or ATM defect Phase 2
Drug: Talazoparib Phase 2 — The dose will be determined after the overall available data (including safety and preliminary anti tumor activity) emerging from the Phase 1b portion of the study have been evaluated.
  Other Names: MDV3800, BMN 673
  Arms: A1. NSCLC Phase 2; A2. NSCLC PD-L1 Resistant DDR+ Phase 2; B1. TNBC Phase 2; B2. HR+BC DDR Defect +Assay Phase 2; C1. Ovarian CA Recurrent Plat-Sensitive Phase 2; C2.Ovarian CA Recurrent Plat-Sensitive BRCA defect Phase 2; D.Urothelial CA Phase 2; E1. CRPC Phase 2; E2. CRPC DDR Defect +Assay Phase 2; F: Advanced Solid Tumors with BRCA or ATM defect Phase 2

SUMMARY:
Avelumab in combination with talazoparib will be investigated in patients with locally advanced (primary or recurrent) or metastatic solid tumors, including non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), hormone receptor positive (HR+) breast cancer, recurrent platinum sensitive ovarian cancer, urothelial cancer (UC), and castration resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
Avelumab is a human immunoglobulin (Ig)G1 monoclonal antibody (mAb) directed against programmed death ligand 1 (PD L1). Avelumab selectively binds to PD L1 and competitively blocks its interaction with programmed death receptor 1 (PD 1), thereby interfering with this key immune checkpoint inhibition pathway. Avelumab is currently being investigated as single agent and in combination with other anti cancer therapies in patients with locally advanced or metastatic solid tumors and various hematological malignancies.

Talazoparib is a potent, orally bioavailable poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor, which is cytotoxic to human cancer cell lines harboring gene mutations that compromise deoxyribonucleic acid (DNA) repair, an effect referred to as synthetic lethality, and by trapping PARP protein on DNA thereby preventing DNA repair, replication, and transcription.

Avelumab in combination with talazoparib will be investigated in patients with locally advanced (primary or recurrent) or metastatic solid tumors, including non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), hormone receptor positive (HR+) breast cancer, recurrent platinum sensitive ovarian cancer, urothelial cancer (UC), and castration resistant prostate cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumors that are not amenable for treatment with curative intent in adult patients with: NSCLC, TNBC, HR+ breast cancer, recurrent platinum sensitive ovarian cancer, UC, CRPC, and other advanced solid tumors with a BRCA or ATM gene defect
* Mandatory primary or metastatic tumor biopsy. If archival tumor tissue is available from a biopsy/surgery the tumor tissue may be submitted without repeating a tumor biopsy during the screening period.
* Minimum age in Japan is 20 years.
* ECOG performance status 0 or 1.
* Resolved acute effects of prior therapy
* Adequate bone marrow, renal, and liver function.
* Negative serum pregnancy test at screening.
* Pregnant, breastfeeding females or female patients able to have children must agree to use highly effective method of contraception throughout the study and for at least 30 days after the last dose of avelumab and for at least 7 months after the last dose of talazoparib; fertile male patients must use a condom during treatment and for at least 4 months after the last dose of talazoparib.
* Signed and dated informed consent.

Exclusion Criteria:

* Prior treatment with a PARP inhibitor.
* Prior immunotherapy with IL-2, IFN-α, or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, OX 40, GITR, LAG 3, IDO, TDO,TIM 3, CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways. Prior treatment with Sipuleucel-T for patients with mCRPC is allowed. For cohort A2 NSCLC patients prior treatment with anti-PD-1/L1 is allowed
* Prior anti-cancer therapy within 2 weeks prior to study enrollment. Prior radiation therapy within 2 weeks prior to enrollment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided it has been completed 2 days prior to study enrollment and no clinically significant toxicities are expected (eg, mucositis, esophagitis).
* Major surgery within 4 weeks prior to study enrollment.
* Current use of immunosuppressive medication at the time of study enrollment.
* Known prior or suspected hypersensitivity to investigational products.
* Known history of immune mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis.
* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Vaccination within 4 weeks of study enrollment and while on trial is prohibited except for administration of inactivated vaccines.
* Diagnosis of Myelodysplastic Syndrome.
* Patients with known brain metastases requiring steroids.
* Participation in other studies involving investigational drug(s) within 4 weeks prior to study participation and/or during study participation.
* Persisting toxicity related to prior therapy >Grade 1
* Known HIV or AIDs-related illness.
* Positive HBV or HCV test indicating acute or chronic infection.
* Active infection requiring systemic therapy.
* Clinically significant cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months prior to study entry; unstable angina, congestive heart failure or a serious cardiac arrhythmia requiring medication.
* Current or anticipated use within 7 days prior to first dose of study drug, or anticipated use during the study of a strong P-gp inhibitor.
* Other acute or chronic medical or psychiatric conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- United States (38):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Highlands Oncology, Springdale, Arkansas
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center/Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Freidenrich Center for Translational Research (CTRU), Palo Alto, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - Stanford Women's Cancer Center, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Massachusetts General Hospital Attn: Lalit Joshi, Boston, Massachusetts
  - Massachusetts General Hospital Attn: Svetlana Rashkova, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Attn: Vasilika Koci, PharmD, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University Of Minesota Health: Clinics And Surgery Center, Minneapolis, Minnesota
  - University of Minesota Medical Center, Fairview IDS Pharmacy, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Roswell Park Cancer Center Institute, Buffalo, New York
  - NYU Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Langone Radiology, New York, New York
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - NYU Langone Radiology - Ambulatory Care Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Hospital- Pharmacy department, New York, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Macquarie University, North Ryde, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Northern Cancer Institute, Sydney, New South Wales
  - Mater Misericordiae Ltd, Brisbane, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Denmark (3):
  - Phase 1 Unit, Department of Oncology, Section 5073., Copenhagen
  - Herlev og Gentofte Hospital, Herlev
  - The Experimental Cancer Therapy Unit, Herlev
- Hungary (3):
  - Orszagos Onkologiai Intezet, Budapest
  - CRU Hungary Kft., Miskolc
  - Pecsi Tudomanyegyetem, Pécs
- Russia (6):
  - Medical Radiological Research Center n.a. A.F. Tsyba -, Obninsk, Kaluga Oblast
  - Medical Radiological Research Center n.a. A.F. Tsyba, Obninsk, Kaluga Oblast
  - GBUZ, Chelyabinsk
  - FSBI "National Medical Research Centre of Oncology n.a., Moscow
  - Budget Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk
  - State budgetary institution of healthcare of Yaroslavl region "Clinical oncology hospital", Yaroslavl
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust, London, Other
  - University Hospitals of Leicester NHS Trust, Leicester
  - Freeman Hospital, The Sir Bobby Robson Cancer Trials, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Yap TA, Bardia A, Dvorkin M, Galsky MD, Beck JT, Wise DR, Karyakin O, Rubovszky G, Kislov N, Rohrberg K, Joy AA, Telli ML, Schram AM, Conte U, Chappey C, Stewart R, Stypinski D, Michelon E, Cesari R, Konstantinopoulos PA. Avelumab Plus Talazoparib in Patients With Advanced Solid Tumors: The JAVELIN PARP Medley Nonrandomized Controlled Trial. JAMA Oncol. 2023 Jan 1;9(1):40-50. doi: 10.1001/jamaoncol.2022.5228. PMID 36394849
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 phases: Phase 1b (talazoparib dose level cohorts) and Phase 2 (expansion phase). The Phase 1b study design started at the highest dose of talazoparib (1 mg QD), to be de-escalated to 0.75 and 0.5 mg QD. With DLT rate <33% among 12 DLT-evaluable patients treated at 1 mg, Phase 2 started. The 2 cohorts at lower dose did not enroll any participants and are not displayed in the results. Only the Phase 1b cohort "Avelumab 800 mg Q2W + Talazoparib 1 mg QD" is displayed.
Pre-assignment Details: Phase 1b: 12 participants were enrolled and assigned to study treatment. Phase 2: 211 participants were enrolled and assigned to study treatment.
Groups:
- Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD: Participants with locally advanced or metastatic solid tumors were treated with talazoparib 1.0 mg orally once daily (QD) in combination with avelumab 800 mg intravenously (IV) every 2 weeks (Q2W) for a maximum of 246.3 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort A1 (NSCLC): Participants with locally advanced (primary or recurrent) or metastatic non-small cell lung cancer (NSCLC) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 183.6 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort A2 (NSCLC DDR+): Participants with locally advanced (primary or recurrent) or metastatic NSCLC with DNA damage repair positive (DDR+) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 173.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort B1 (TNBC): Participants with locally advanced (primary or recurrent) or triple-negative breast cancer (TNBC) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 93.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort B2 (BC HR+ HER2- DDR+): Participants with locally advanced (primary or recurrent) or metastatic hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer (BC) with DDR+ were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 180.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort C1 (OVC): Participants with locally advanced (primary or recurrent) or metastatic ovarian cancer (OVC) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 161.1 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort C2 (OVC BRCA-mutated): Participants with locally advanced (primary or recurrent) or metastatic OVC with germline or somatic BRCA1 or BRCA2 gene defect were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 144.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort D (UC): Participants with locally advanced (primary or recurrent) or metastatic urothelial cancer (UC) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 164.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort E1 (mCRPC): Participants with metastatic castration-resistant prostate cancer (mCRPC) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 54.1 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort E2 (mCRPC DDR+): Participants with mCRPC with DDR+ were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 74.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort F (BRCA/ATM-mutated): Participants with locally advanced (primary or recurrent) or metastatic solid tumors, independent of tissue of origin, with previously identified pathogenic, or likely pathogenic, germline or somatic defects in BRCA1, BRCA2, or ATM genes were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 49.9 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Period: Overall Study
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Started | 12 | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Not completed — Other | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 8 | 27 | 4 | 18 | 16 | 14 | 7 | 29 | 9 | 11 | 5
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 1
Not completed — Global deterioration of health status | 2 | 3 | 0 | 2 | 3 | 3 | 0 | 2 | 8 | 4 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 4 | 2 | 2 | 2
Not completed — Death | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated) | Total
Number analyzed (Participants) | 12 | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9 | 223
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 62.67 (9.49) | 67.00 (9.37) | 59.60 (7.40) | 56.18 (12.49) | 53.83 (14.08) | 62.65 (10.66) | 61.36 (9.24) | 65.73 (9.19) | 63.71 (7.40) | 71.56 (7.37) | 63.00 (10.91) | 63.17 (11.04)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 6 | 15 | 4 | 15 | 17 | 12 | 7 | 16 | 8 | 3 | 5 | 108
  65 - <75 years | 5 | 19 | 1 | 6 | 3 | 5 | 3 | 16 | 12 | 8 | 2 | 80
  75 - <85 years | 1 | 7 | 0 | 1 | 3 | 3 | 1 | 7 | 1 | 6 | 2 | 32
  >= 85 years | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 2 | 22 | 22 | 20 | 11 | 14 | 0 | 0 | 3 | 106
  Male | 9 | 33 | 3 | 0 | 1 | 0 | 0 | 26 | 21 | 18 | 6 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 7
  Not Hispanic or Latino | 12 | 39 | 5 | 19 | 21 | 18 | 11 | 38 | 11 | 16 | 8 | 198
  Unknown or Not Reported | 0 | 3 | 0 | 3 | 1 | 2 | 0 | 0 | 7 | 1 | 1 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 2 | 0 | 14
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 5 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 2 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 9 | 34 | 4 | 20 | 17 | 18 | 6 | 36 | 12 | 14 | 9 | 179
  Not reported | 0 | 2 | 0 | 1 | 4 | 2 | 0 | 1 | 3 | 0 | 0 | 13
Geographic Region [Count of Participants; unit: Participants]
  North America | 12 | 9 | 3 | 14 | 15 | 10 | 7 | 15 | 20 | 11 | 8 | 124
  Western Europe | 0 | 10 | 2 | 0 | 1 | 2 | 1 | 5 | 1 | 4 | 1 | 27
  Eastern Europe | 0 | 19 | 0 | 6 | 4 | 5 | 1 | 16 | 0 | 1 | 0 | 52
  Australasia | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 10
  Asia | 0 | 4 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 10
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG=Eastern Cooperative Oncology Group. Score 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work or office work.
  Participants
    0 | 4 | 5 | 1 | 12 | 12 | 9 | 8 | 16 | 4 | 6 | 1 | 78
    1 | 8 | 37 | 4 | 10 | 11 | 11 | 3 | 24 | 17 | 12 | 8 | 145

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs=occurrence of any of the following AEs attributable to any study treatment in Cycle 1:Hematologic: grade(G)4 neutropenia lasting >5 days (absolute neutrophil count [ANC]< 0.5*10^9/L); febrile neutropenia; neutropenic infection (ANC<1.0*10^9/L, and G>3 infection); G>=3 thrombocytopenia (platelet count [PC] <50.0*10^9/L) with bleeding; G4 thrombocytopenia (PC<25.0*10^9/L); G4 anemia (life-threatening; urgent intervention indicated). Non-hematologic: G>=3 toxicities unless predefined in the protocol; potential Hy's law cases. Non-adherence to treatment schedule: failure to deliver at least 75% of the planned doses of talazoparib during the first cycle of treatment due to treatment-related toxicities; G3 non-hematologic toxicity that delayed administration of either study drug for more than 2 weeks. Dose reductions: any adverse event (AE) that resulted in a dose reduction of talazoparib.
Time Frame: Cycle 1; 28 days
Population: The DLT analysis set was a subset of the safety analysis set and included all enrolled participants in the Phase 1b portion who were eligible for the study, received at least 1 dose of the combination treatment, and either experienced DLT during the first cycle (28 days) of treatment, or completed the DLT observation period for the first cycle of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD: Participants with locally advanced or metastatic solid tumors were treated with talazoparib 1.0 mg orally QD in combination with avelumab 800 mg IV Q2W for a maximum of 246.3 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 12
Participants | 3

2. Primary Outcome: Phase 2: Percentage of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 by Investigator Assessment
Description: This outcome measure (OM) is reported for participants with solid tumors except mCRPC; for those participants, OR was defined as a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors (RECIST) version(v) 1.1 by investigator. CR: Complete disappearance of all target and non-target lesions with the exception of nodal disease; all target and non-target nodes must decrease to normal size (short axis <10 mm); all lesions must be assessed. PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions; all target lesions must be assessed. Non-target PR lesions must be non-progressive disease (PD), where PD is unequivocal progression of pre-existing lesions.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 4.3 years approximately)
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was not planned to be collected and analyzed for Phase 1b arm. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 2: Cohort A2 (NSCLC DDR+): Participants with locally advanced (primary or recurrent) or metastatic NSCLC with DNA damage repair positive (DDR+) were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 183.6 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
- Phase 2: Cohort B2 (BC HR+ HER2- DDR+): Participants with locally advanced (primary or recurrent) or metastatic hormone receptor positive (HR+)/herman epidermal growth factor receptor 2 negative (HER2-) breast cancer (BC) with DDR+ were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 180.0 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 7
Percentage of Participants | 16.7 [7.0 to 31.4] | 20.0 [0.5 to 71.6] | 18.2 [5.2 to 40.3] | 34.8 [16.4 to 57.3] | 20.0 [5.7 to 43.7] | 63.6 [30.8 to 89.1] | 15.0 [5.7 to 29.8] | 0 [0.0 to 41.0]

3. Primary Outcome: Phase 2: Percentage of Participants With Confirmed Objective Response (OR) as Per RECIST v1.1 and Prostate Cancer Working Group 3 (PCWG3) by Investigator Assessment
Description: This OM is reported for participants with mCRPC; for those participants, OR was defined as the proportion of participants with a best overall soft tissue response of CR or PR per RECIST v1.1 and with no evidence of confirmed bone disease progression per PCWG3 criteria by investigator. CR: Complete disappearance of all target and non-target lesions with the exception of nodal disease; all target and non-target nodes must decrease to normal size (short axis <10 mm); all lesions must be assessed. PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions; all target lesions must be assessed. Non-target PR lesions must be non-PD.
Time Frame: as for outcome 2
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was not planned to be collected and analyzed for Phase 1b arm. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 21 | 18 | 2
Percentage of Participants | 0 [0.0 to 16.1] | 11.1 [1.4 to 34.7] | 50.0 [1.3 to 98.7]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received any study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs).
Time Frame: From start of the treatment up to 30 days after last dose or start of new anticancer therapy minus 1 day, whichever occurred first (maximum up to 5.2 years approximately)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug. Cohorts in Phase 2 were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: All participants from Cohort A to Cohort F combined.
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality TEAEs | 12 | 207
  Participants with treatment-related TEAEs | 11 | 197

5. Secondary Outcome: Number of Participants With Grade >=3 TEAEs
Description: AE was any untoward medical occurrence in a participant who received any study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. TEAEs were graded by the investigator using National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v 4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. In this outcome measure, number of participants with Grade 3 or higher TEAEs were reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality Grade >=3 TEAEs | 9 | 156
  Participants with treatment-related Grade >=3 TEAEs | 9 | 120

6. Secondary Outcome: Number of Participants With Serious TEAEs
Description: TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs). A serious TEAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/considered to be an important medical event: death; life-threatening experience (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality serious TEAEs | 1 | 75
  Participants with treatment-related serious TEAEs | 1 | 25

7. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation of Either Study Drug
Description: Either study drug = avelumab only or talazoparib only. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality TEAEs leading to discontinuation of avelumab only | 0 | 5
  Participants with treatment-related TEAEs leading to discontinuation of avelumab only | 0 | 4
  Participants with all-causality TEAEs leading to discontinuation of talazoparib only | 1 | 9
  Participants with treatment-related TEAEs leading to discontinuation of talazoparib only | 1 | 8

8. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation of All Study Drugs
Description: All study drugs = all study drugs in the combination. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality TEAEs leading to discontinuation of all study drugs | 1 | 20
  Participants with treatment-related TEAEs leading to discontinuation of all study drugs | 0 | 1

9. Secondary Outcome: Number of Participants With TEAEs Leading to Death
Description: TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Participants with all-causality TEAEs leading to death | 0 | 21
  Participants with treatment-related TEAEs leading to death | 0 | 1

10. Secondary Outcome: Number of Participants With New or Worsening Hematology Laboratory Test Results to Grade >=1 During the On-Treatment Period
Description: The number of participants with newly occurring or worsening hematology abnormalities during the on-treatment period were summarized by worst grade on-treatment. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. NCI-CTCAE criteria version 4.03 is used. As per NCI CTCAE toxicity grading v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
Time Frame: as for outcome 4
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug. Cohorts in Phase 2 were combined as pre-specified in reporting and analysis plan. Here 'number analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD: Participants with locally advanced or metastatic solid tumors were treated with talazoparib 1.0 mg orally QD in combination with avelumab 800 mg IV Q2W for a maximum of246.3 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 11 | 143
  Activated partial thromboplastin time prolonged | 4 | 21
  Anemia: number analyzed (Participants) | 12 | 208
  Anemia | 8 | 161
  Hemoglobin increased: number analyzed (Participants) | 12 | 208
  Hemoglobin increased | 0 | 1
  Lymphocyte count decreased: number analyzed (Participants) | 12 | 208
  Lymphocyte count decreased | 9 | 145
  Lymphocyte count increased: number analyzed (Participants) | 12 | 208
  Lymphocyte count increased | 1 | 3
  Neutrophil count decreased: number analyzed (Participants) | 12 | 208
  Neutrophil count decreased | 8 | 100
  Platelet count decreased: number analyzed (Participants) | 12 | 208
  Platelet count decreased | 6 | 141
  White blood cell decreased: number analyzed (Participants) | 12 | 208
  White blood cell decreased | 10 | 139

11. Secondary Outcome: Number of Participants With New or Worsening Hematology Laboratory Test Results to Grade >=3 During the On-Treatment Period
Description: as for outcome 10
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 11 | 143
  Activated partial thromboplastin time prolonged | 0 | 1
  Anemia: number analyzed (Participants) | 12 | 208
  Anemia | 4 | 78
  Lymphocyte count decreased: number analyzed (Participants) | 12 | 208
  Lymphocyte count decreased | 4 | 44
  Neutrophil count decreased: number analyzed (Participants) | 12 | 208
  Neutrophil count decreased | 5 | 27
  Platelet count decreased: number analyzed (Participants) | 12 | 208
  Platelet count decreased | 4 | 47
  White blood cell decreased: number analyzed (Participants) | 12 | 208
  White blood cell decreased | 3 | 20

12. Secondary Outcome: Number of Participants With New or Worsening Chemistry Laboratory Test Results to Grade >=1 During the On-Treatment Period
Description: The number of participants with newly occurring or worsening chemistry abnormalities during the on-treatment period were summarized by worst grade on-treatment. On-treatment period was defined as time from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. NCI-CTCAE criteria version 4.03 is used. As per NCI CTCAE toxicity grading v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Alanine aminotransferase increased: number analyzed (Participants) | 12 | 208
  Alanine aminotransferase increased | 1 | 41
  Alkaline phosphatase increased: number analyzed (Participants) | 12 | 208
  Alkaline phosphatase increased | 3 | 74
  Aspartate aminotransferase increased: number analyzed (Participants) | 12 | 208
  Aspartate aminotransferase increased | 2 | 53
  Blood bilirubin increased: number analyzed (Participants) | 12 | 208
  Blood bilirubin increased | 0 | 24
  Creatinine Phosphokinase (CPK) increased: number analyzed (Participants) | 12 | 206
  Creatinine Phosphokinase (CPK) increased | 2 | 37
  Creatinine increased: number analyzed (Participants) | 12 | 208
  Creatinine increased | 9 | 147
  Gamma-glutamyl transferase (GGT) increased: number analyzed (Participants) | 12 | 206
  Gamma-glutamyl transferase (GGT) increased | 2 | 69
  Hypercalcemia: number analyzed (Participants) | 12 | 208
  Hypercalcemia | 1 | 23
  Hyperglycemia: number analyzed (Participants) | 12 | 208
  Hyperglycemia | 0 | 48
  Hyperkalemia: number analyzed (Participants) | 12 | 208
  Hyperkalemia | 2 | 25
  Hypermagnesemia: number analyzed (Participants) | 12 | 207
  Hypermagnesemia | 0 | 21
  Hypernatremia: number analyzed (Participants) | 12 | 208
  Hypernatremia | 0 | 9
  Hypoalbuminemia: number analyzed (Participants) | 12 | 208
  Hypoalbuminemia | 2 | 60
  Hypocalcemia: number analyzed (Participants) | 12 | 208
  Hypocalcemia | 1 | 45
  Hypoglycemia: number analyzed (Participants) | 12 | 208
  Hypoglycemia | 0 | 13
  Hypokalemia: number analyzed (Participants) | 12 | 208
  Hypokalemia | 3 | 36
  Hypomagnesemia: number analyzed (Participants) | 12 | 207
  Hypomagnesemia | 2 | 33
  Hyponatremia: number analyzed (Participants) | 12 | 208
  Hyponatremia | 4 | 66
  Hypophosphatemia: number analyzed (Participants) | 12 | 206
  Hypophosphatemia | 2 | 43
  Lipase increased: number analyzed (Participants) | 12 | 207
  Lipase increased | 4 | 36
  Serum amylase increased: number analyzed (Participants) | 12 | 207
  Serum amylase increased | 2 | 32

13. Secondary Outcome: Number of Participants With New or Worsening Chemistry Laboratory Test Results to Grade >=3 During the On-Treatment Period
Description: as for outcome 12
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  Alanine aminotransferase increased: number analyzed (Participants) | 12 | 208
  Alanine aminotransferase increased | 0 | 2
  Alkaline phosphatase increased: number analyzed (Participants) | 12 | 208
  Alkaline phosphatase increased | 0 | 7
  Aspartate aminotransferase increased: number analyzed (Participants) | 12 | 208
  Aspartate aminotransferase increased | 0 | 2
  Blood bilirubin increased: number analyzed (Participants) | 12 | 208
  Blood bilirubin increased | 0 | 3
  Creatinine Phosphokinase (CPK) increased: number analyzed (Participants) | 12 | 206
  Creatinine Phosphokinase (CPK) increased | 0 | 4
  Creatinine increased: number analyzed (Participants) | 12 | 208
  Creatinine increased | 0 | 2
  Gamma-glutamyl transferase (GGT) increased: number analyzed (Participants) | 12 | 206
  Gamma-glutamyl transferase (GGT) increased | 0 | 11
  Hyperglycemia: number analyzed (Participants) | 12 | 208
  Hyperglycemia | 0 | 6
  Hyperkalemia: number analyzed (Participants) | 12 | 208
  Hyperkalemia | 0 | 1
  Hypermagnesemia: number analyzed (Participants) | 12 | 207
  Hypermagnesemia | 0 | 5
  Hypoalbuminemia: number analyzed (Participants) | 12 | 208
  Hypoalbuminemia | 0 | 2
  Hypocalcemia: number analyzed (Participants) | 12 | 208
  Hypocalcemia | 0 | 4
  Hypokalemia: number analyzed (Participants) | 12 | 208
  Hypokalemia | 0 | 1
  Hyponatremia: number analyzed (Participants) | 12 | 208
  Hyponatremia | 0 | 12
  Hypophosphatemia: number analyzed (Participants) | 12 | 206
  Hypophosphatemia | 1 | 6
  Lipase increased: number analyzed (Participants) | 12 | 207
  Lipase increased | 0 | 14
  Serum amylase increased: number analyzed (Participants) | 12 | 207
  Serum amylase increased | 0 | 7

14. Secondary Outcome: Trough Concentrations (Ctrough)/Predose and Maximum Concentrations (Cmax) of Serum Avelumab Concentrations (μg/mL) by Visit (Excluding Site 1055)
Description: Pharmacokinetics (PK) data analyses included descriptive summary statistics of the pre-dose/Ctrough concentrations for both investigational products and post-dose (for talazoparib) or Cmax concentrations (for avelumab) for each cycle.
Time Frame: Predose/0 Hour (H) and 1 H on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2-4, and additionally on Day 1 of Cycles 6, 9, 12, 18, and 24.
Population: The PK concentration analysis sets (1 unique set for each study drug used in the combination) were subsets of safety analysis set including participants with >=1 post-dose concentration measurement above the lower limit of quantitation (LLQ) for avelumab/talazoparib. Cohorts were combined as pre-specified in reporting and analysis plan. Site 1055 was excluded as samples were not meeting the protocol requirements. Here 'number analyzed' signifies participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Phase 1b and Phase 2 Combined: Treatment = Avelumab 800 mg IV Infusion Q2W coadministered with Talazoparib 1 mg QD.
Arm/Group | Phase 1b and Phase 2 Combined
Number analyzed (Participants) | 194
μg/mL
  Cycle 1 / Day 1 (0 Hour [H]) | NA (NA) — The result was Not Available as no observations were above the avelumab LLQ of 0.2 μg/mL.
  Cycle 1 / Day 1 (1 H): number analyzed (Participants) | 178
  Cycle 1 / Day 1 (1 H) | 221.0 (41)
  Cycle 1 / Day 15 (0 H): number analyzed (Participants) | 183
  Cycle 1 / Day 15 (0 H) | 21.20 (72)
  Cycle 1 / Day 15 (1 H): number analyzed (Participants) | 164
  Cycle 1 / Day 15 (1 H) | 206.6 (86)
  Cycle 2 / Day 1 (0 H): number analyzed (Participants) | 168
  Cycle 2 / Day 1 (0 H) | 26.41 (68)
  Cycle 2 / Day 1 (1 H): number analyzed (Participants) | 156
  Cycle 2 / Day 1 (1 H) | 199.6 (110)
  Cycle 3 / Day 1 (0 H): number analyzed (Participants) | 120
  Cycle 3 / Day 1 (0 H) | 31.45 (80)
  Cycle 3 / Day 1 (1 H): number analyzed (Participants) | 126
  Cycle 3 / Day 1 (1 H) | 188.8 (105)
  Cycle 4 / Day 1 (0 H): number analyzed (Participants) | 106
  Cycle 4 / Day 1 (0 H) | 34.59 (81)
  Cycle 4 / Day 1 (1 H): number analyzed (Participants) | 114
  Cycle 4 / Day 1 (1 H) | 190.6 (99)
  Cycle 6 / Day 1 (0 H): number analyzed (Participants) | 78
  Cycle 6 / Day 1 (0 H) | 37.40 (73)
  Cycle 6 / Day 1 (1 H): number analyzed (Participants) | 81
  Cycle 6 / Day 1 (1 H) | 185.9 (98)
  Cycle 9 / Day 1 (0 H): number analyzed (Participants) | 40
  Cycle 9 / Day 1 (0 H) | 39.97 (91)
  Cycle 9 / Day 1 (1 H): number analyzed (Participants) | 44
  Cycle 9 / Day 1 (1 H) | 171.1 (145)
  Cycle 12 / Day 1 (0 H): number analyzed (Participants) | 18
  Cycle 12 / Day 1 (0 H) | 47.10 (63)
  Cycle 12 / Day 1 (1 H): number analyzed (Participants) | 18
  Cycle 12 / Day 1 (1 H) | 202.9 (88)
  Cycle 18 / Day 1 (0 H): number analyzed (Participants) | 3
  Cycle 18 / Day 1 (0 H) | 53.94 (33)
  Cycle 18 / Day 1 (1 H): number analyzed (Participants) | 3
  Cycle 18 / Day 1 (1 H) | 135.6 (354)
  Cycle 24 / Day 1 (0 H): number analyzed (Participants) | 1
  Cycle 24 / Day 1 (0 H) | 76.40 (NA) — Only 1 participant evaluable for this timepoint. Coefficient of variation is not applicable.
  Cycle 24 / Day 1 (1 H): number analyzed (Participants) | 1
  Cycle 24 / Day 1 (1 H) | 378.0 (NA) — Only 1 participant evaluable for this timepoint. Coefficient of variation is not applicable.

15. Secondary Outcome: Predose and Postdose Plasma Talazoparib Concentrations (pg/mL) by Visit (Excluding Site 1055)
Description: Pharmacokinetics (PK) data analyses included descriptive summary statistics of the pre-dose/Ctrough concentrations for both investigational products and post-dose (for talazoparib) or Cmax concentrations (for avelumab) for each cycle. Cmax=maximum concentration. Ctrough=trough concentration. Participants with moderate renal impairment were started at a lower, 0.75 mg QD, dose to compensate for decreased talazoparib clearance.
Time Frame: Pre-dose and post-dose (at the end of the avelumab infusion) on Days 1 and 15 of Cycle 1 and on Day 1 of Cycles 2-4.
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Talazoparib Starting Dose = 1 mg QD: Treatment = Avelumab 800 mg IV Infusion Q2W coadministered with Talazoparib 1 mg QD (participants with normal renal function or mild renal impairment).
- Talazoparib Starting Dose = 0.75 mg QD: Treatment = Avelumab 800 mg IV Infusion Q2W coadministered with Talazoparib 0.75 mg QD (participants with moderate renal impairment)
Arm/Group | Talazoparib Starting Dose = 1 mg QD | Talazoparib Starting Dose = 0.75 mg QD
Number analyzed (Participants) | 163 | 31
pg/mL
  Cycle 1 / Day 1 (Predose) | NA (NA) — The result was Not Available as no observations were above the talazoparib LLQ of 25 pg/mL. | NA (NA) — The result was Not Available as no observations were above the talazoparib LLQ of 25 pg/mL.
  Cycle 1 / Day 1 (Postdose): number analyzed (Participants) | 46 | 12
  Cycle 1 / Day 1 (Postdose) | 2295 (137) | 2015 (112)
  Cycle 1 / Day 15 (Predose): number analyzed (Participants) | 72 | 10
  Cycle 1 / Day 15 (Predose) | 4672 (63) | 4657 (47)
  Cycle 1 / Day 15 (Postdose): number analyzed (Participants) | 33 | 3
  Cycle 1 / Day 15 (Postdose) | 9055 (88) | 8257 (11)
  Cycle 2 / Day 1 (Predose): number analyzed (Participants) | 66 | 10
  Cycle 2 / Day 1 (Predose) | 4385 (53) | 5871 (53)
  Cycle 2 / Day 1 (Postdose): number analyzed (Participants) | 21 | 5
  Cycle 2 / Day 1 (Postdose) | 8479 (73) | 9834 (62)
  Cycle 3 / Day 1 (Predose): number analyzed (Participants) | 47 | 6
  Cycle 3 / Day 1 (Predose) | 4212 (46) | 3874 (48)
  Cycle 3 / Day 1 (Postdose): number analyzed (Participants) | 22 | 3
  Cycle 3 / Day 1 (Postdose) | 6765 (239) | 1236 (8074)
  Cycle 4 / Day 1 (Predose): number analyzed (Participants) | 29 | 6
  Cycle 4 / Day 1 (Predose) | 4713 (38) | 3826 (73)
  Cycle 4 / Day 1 (Postdose): number analyzed (Participants) | 15 | 3
  Cycle 4 / Day 1 (Postdose) | 6506 (76) | 6735 (70)

16. Secondary Outcome: Number of Participants With at Least 1 Valid Anti-drug Antibody (ADA) Result at: Any Time Point (N0), Baseline (N1), Baseline and Post-Baseline (N2), and Post-Baseline and Without Positive Baseline ADA Result (N3)
Description: Immunogenicity blood samples were assayed for ADA using a validated assay. The sample analysis followed a tiered approach of screening, confirmation, and titer determination. Samples tested positive for ADA were further analyzed for neutralizing antibodies (Nab) using a validated assay. Baseline was defined as the last assessment prior to the date/time of the first dose of avelumab. N0, N1, N2, and N3=Number of participants with at least 1 valid ADA result at any time point, baseline (pre-dose on Day 1), baseline and post-baseline, and post-baseline, respectively.
Time Frame: Pre-dose (within 2 hours of talazoparib dose) on Day 1 and Day 15 of Cycle 1, on Day 1 of Cycle 2-4 and then on Day 1 of Cycles 6, 9, 12, 18, 24, and at the end of treatment (EOT)
Population: The immunogenicity analysis set was a subset of the safety analysis set and included participants who had at least 1 ADA/Nab sample collected for avelumab. Cohorts in Phase 2 were combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  N0 | 12 | 211
  N1 | 12 | 209
  N2 | 11 | 202
  N3 | 11 | 200

17. Secondary Outcome: Number of Participants by ADA Categories
Description: Immunogenicity blood samples were assayed for ADA using a validated assay. The sample analysis followed a tiered approach of screening, confirmation, and titer determination. Samples tested positive for ADA were further analyzed for neutralizing antibodies (Nab) using a validated assay. Baseline was defined as the last assessment prior to the date/time of the first dose of avelumab. N0, N1, N2, and N3=Number of participants with at least 1 valid ADA Result at any time point, baseline (pre-dose on Day 1), baseline and post-baseline, and post-baseline, respectively. n=number of participants in each category.
Time Frame: Pre-dose (within 2 hours of talazoparib dose) on Day 1 and Day 15 of Cycles 1, on Day 1 of Cycle 2-4 and then on Day 1 of Cycles 6, 9, 12, 18, 24, and at the end of treatment (EOT)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2
Number analyzed (Participants) | 12 | 211
Participants
  ADA never-positive (n/N0) | 12 | 205
  ADA ever-positive (n/N0) | 0 | 6
  ADA ever-positive: Baseline ADA positive (n/N1) (No treatment-boosted ADA [n/N2]) | 0 | 4
  ADA ever-positive: Treatment-induced ADA positive (n/N3) | 0 | 2

18. Secondary Outcome: Phase 1b: Percentage of Participants With Confirmed OR as Per RECIST v1.1 and PCWG3 by Investigator Assessment
Description: This OM is reported for participants in Phase 1b; OR was defined as the proportion of participants with a best overall soft tissue response of CR or PR per RECIST v1.1 and with no evidence of confirmed bone disease progression per Prostate Cancer Working Group 3 (PCWG3) criteria by investigator. CR: Complete disappearance of all target and non-target lesions with the exception of nodal disease; all target and non-target nodes must decrease to normal size (short axis <10 mm); all lesions must be assessed. PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions; all target lesions must be assessed. Non-target PR lesions must be non-PD.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 1b arm only.
Measure: Number (95% Confidence Interval); unit: Percentage of Particpants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 12
Percentage of Particpants | 16.7 [2.1 to 48.4]

19. Secondary Outcome: Phase 1b: Time to Response (TTR) in Participants With Confirmed CR or PR
Description: For participants with solid tumors except mCRPC, TTR was defined for participants with confirmed OR (CR or PR) as the time from the first dose of study treatment to the first documentation of objective tumor response. For participants with mCRPC, TTR was defined as the time from the first dose of study treatment to the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression on bone scan per PCWG3. Soft tissue response was defined as a best overall response (BOR) of CR or PR as assessed by Investigator using RECIST v1.1.
Time Frame: From the first dose of study treatment to the first documentation of objective tumor response/the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression (<=5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 1b arm only. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 2
Months | 1.8 [1.8 to 1.8]

20. Secondary Outcome: Phase 2: TTR in Participants With Confirmed CR or PR
Description: as for outcome 19
Time Frame: From the first dose of study treatment to the first documentation of objective tumor response/the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression (<= 5.2 years approximately)
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 2 only. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 7 | 1 | 4 | 8 | 4 | 7 | 6 | 2 | 1
Months | 3.7 [1.7 to 11.3] | 1.8 [1.8 to 1.8] | 1.8 [1.6 to 2.0] | 1.9 [1.6 to 3.6] | 3.6 [1.7 to 17.9] | 1.7 [1.6 to 3.7] | 2.1 [1.4 to 5.9] | 5.5 [5.4 to 5.6] | 1.8 [1.8 to 1.8]

21. Secondary Outcome: Phase 2: Duration of Response (DR) in Participants With Confirmed CR or PR
Description: For participants with solid tumors except mCRPC, DR was defined for participants with confirmed OR (CR or PR) as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first.
Time Frame: From the first objective tumor response/soft tissue response to the first objective tumor progression/subsequent objective evidence of radiographic progression or death due to any cause, whichever occurred first (<=5.2 years approximately)
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 2 only. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure; Cohorts without evaluable participants for this outcome measure [i.e., Phase 2: Cohort E1 (mCRPC), Phase 2: Cohort E2 (mCRPC DDR+), Phase 2: Cohort F (BRCA/ATM-mutated)] are not presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC)
Number analyzed (Participants) | 7 | 1 | 4 | 8 | 4 | 7 | 6
Months | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants | NA [NA to NA] — Median and 95% CI were not estimated for <10 participants

22. Secondary Outcome: Phase 1b: Progression-Free Survival (PFS) in Participants With Confirmed CR or PR
Description: For participants with solid tumors except mCRPC, PFS was defined as the time from the first dose of study treatment to the date of disease progression by RECIST v1.1 or death due to any cause, whichever occurred first. For participants with mCRPC, PFS was defined as the time from the first dose of study treatment to documentation of radiographic progression in soft tissue as assessed by Investigator using RECIST v1.1, in bone as assessed by Investigator using PCWG3, or death, whichever occurred first
Time Frame: From the first dose of study treatment to the date of disease progression/radiographic progression in soft tissue or bone, or death due to any cause, whichever occurred first (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 1b only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 12
Months | 6.0 [1.8 to 11.5]

23. Secondary Outcome: Phase 2: PFS in Participants With Confirmed CR or PR (RECIST v1.1)
Description: This OM is reported for participants with solid tumors except mCRPC; for those participants, PFS was defined as the time from the first dose of study treatment to the date of disease progression by RECIST v1.1 or death due to any cause, whichever occurred first.
Time Frame: as for outcome 22
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 7
Months | 4.7 [3.7 to 7.4] | 1.9 [1.8 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 3.6 [1.9 to 5.6] | 5.3 [2.0 to 12.8] | 7.2 [4.0 to 9.1] | 16.8 [7.2 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 3.6 [1.9 to 5.4] | 1.7 [1.4 to 3.3]

24. Secondary Outcome: Phase 2: PFS in Participants With Confirmed CR or PR (RECIST v1.1 and PCWG3)
Description: This OM was reported for participants with mCRPC; for these participants, PFS was defined as the time from the first dose of study treatment to documentation of radiographic progression in soft tissue as assessed by Investigator using RECIST v1.1, in bone as assessed by Investigator using PCWG3, or death, whichever occurred first.
Time Frame: as for outcome 22
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Phase 2 only. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 21 | 18 | 2
Months | 4.1 [1.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 4.6 [1.7 to 9.8] | 8.4 [5.9 to 10.9]

25. Secondary Outcome: Phase 2: Time to Prostate-Specific Antigen (PSA) Progression for Participants With mCRPC
Description: Time to PSA progression for participants with mCRPC was defined as the time from the first dose to the date that a >=25% increase in PSA with an absolute increase of >=2 μg/L (2 ng/mL) above the nadir (or baseline for participants with no PSA decline) was documented, confirmed by a second consecutive PSA value obtained >=3 weeks (21 days) later.
Time Frame: From the first dose to the date that a >=25% increase in PSA with an absolute increase of >=2 μg/L (2 ng/mL) above the nadir (or baseline for participants with no PSA decline) was documented (maximum up to 5.2 years approximately)
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2: Cohort E2 (mCRPC DDR+): Participants with mCRPC with DDR+ were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 74.1 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 21 | 18 | 2
Months | 1.0 [1.0 to 4.6] | 2.8 [1.0 to 6.5] | 3.1 [1.6 to 4.6]

26. Secondary Outcome: Phase 1b: Overall Survival
Description: Overall survival (OS) was defined as the time from the first dose of study treatment to the date of death. Participants without an event (death) were censored at the date of last contact.
Time Frame: From the first dose of study treatment to the date of death (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was for Phase 1b only.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD: Participants with locally advanced or metastatic solid tumors were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 246.3 weeks. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 12
Months | 18.5 [6.4 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event.

27. Secondary Outcome: Phase 2: Overall Survival
Description: OS was defined as the time from the first dose of study treatment to the date of death. Participants without an event (death) were censored at the date of last contact.
Time Frame: From the first dose of study treatment to the date of death (maximum up to 5.2 years approximately)
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was for Phase 2 only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Months | 11.6 [8.4 to 14.9] | 26.3 [3.5 to 43.3] | 8.2 [5.8 to 13.0] | 27.5 [12.6 to 40.2] | 22.9 [7.8 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 38.8 [16.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 13.1 [8.5 to 19.2] | 15.9 [9.6 to 20.7] | 16.1 [10.8 to 23.4] | 6.9 [1.4 to 27.4]

28. Secondary Outcome: Phase 2: Percentage of Participants With PSA Response
Description: PSA response was defined as the proportion of participants with confirmed PSA decline >=50% compared to baseline. PSA response was calculated as a decline from baseline PSA (ng/mL) to the maximal PSA response with a threshold of 50%. A PSA response must be confirmed by a second consecutive value at least 3 weeks later.
Time Frame: From baseline PSA (ng/mL) to the maximal PSA response with a threshold of 50% (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was planned for Cohorts E1, E2, and F in Phase 2 only as pre-specified in reporting and analysis plan. Cohorts without evaluable participants for this outcome measure [ie, Phase 2: Cohort F (BRCA/ATM-mutated)] are not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+)
Number analyzed (Participants) | 21 | 18
Percentage of Participants | 9.5 [1.2 to 30.4] | 5.6 [0.1 to 27.3]

29. Secondary Outcome: Phase 1b: Percentage of Participants With CA-125 Response
Description: Cancer Antigen 125 (CA-125) response is defined as at least a 50% reduction in CA-125 levels from baseline. The response must be confirmed and maintained for at least 28 days.
Time Frame: From baseline to at least a 50% reduction in CA-125 level (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was for Phase 1b only. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD
Number analyzed (Participants) | 1
Percentage of Participants | 100 [2.5 to 100.0]

30. Secondary Outcome: Phase 2: Percentage of Participants With CA-125 Response
Description: CA-125 response is defined as at least a 50% reduction in CA-125 levels from baseline. The response must be confirmed and maintained for at least 28 days.
Time Frame: From baseline to at least a 50% reduction in CA-125 level (maximum up to 5.2 years approximately)
Population: The FAS included all enrolled participants who received at least 1 dose of study treatment. Data for this OM was for Cohorts C1 and C2 in Phase 2 only as pre-specified in reporting and analysis plan.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 2: Cohort C2 (OVC BRCA-mutated): Participants with locally advanced (primary or recurrent) or metastatic OVC with germline or somatic BRCA1 or BRCA2 gene defect were treated with talazoparib 1 mg QD orally in combination with avelumab 800 mg IV Q2W for a maximum of 144.0. Safety follow-up was for 90 days after last dose of study treatment or until time of initiation of new anticancer treatment, whichever comes first.
Arm/Group | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated)
Number analyzed (Participants) | 20 | 11
Percentage of Participants | 45.0 [23.1 to 68.5] | 63.6 [30.8 to 89.1]

31. Secondary Outcome: Number of Participants With Different Programmed Death-Ligand 1 (PD-L1) Status at Baseline
Description: PD-L1 expression on tumor and infiltrating immune cells were measured by immunohistochemistry (IHC). PD-L1 expression level corresponds to the percentage of positive cells. The PD-L1 Positive category does not apply to cohorts A1 and A2. The PD-L1 High/Low categories only apply to cohorts A1 and A2. Participants were considered positive if their baseline tumor tissue sample demonstrated cell surface PD-L1 expression: 1) for Cohorts E1, E2, and F: >=1% tumor cells (TC) or >= 5% immune cells (IC); 2) for Cohort D: TC/IC>=25%; 3) for Cohorts B1, B2, C1, C2: IC>=5%; otherwise were considered negative. Categories based on PD-L1 expression level ≥50% and <50% were defined as High and Low, respectively.
Time Frame: At baseline (the last available assessment prior to the start of study treatment was defined as 'baseline' value or 'baseline' assessment)
Population: The full analysis set (FAS) included all enrolled participants who received at least 1 dose of study treatment. Data for this outcome measure was presented for Phase 2 only as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Participants
  High | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Low | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Positive (Not applicable for Cohorts A1 and A2) | 0 | 0 | 8 | 3 | 5 | 5 | 13 | 1 | 2 | 0
  Negative | 22 | 2 | 6 | 16 | 13 | 4 | 19 | 13 | 12 | 3
  Unknown | 9 | 1 | 8 | 4 | 2 | 2 | 8 | 7 | 4 | 6

32. Secondary Outcome: Number of Participants With Different Tumor Mutational Burden (TMB) at Baseline
Description: TMB was defined as the total number of mutations in the tumor genome, or number of mutations per megabase of DNA if derived from targeted sequencing. High: TMB score >=20 muts/mb (number of mutations per megabase of DNA); Medium: TMB score >=10 muts/mb and <20 muts/mb; Low: TMB score <10 muts/mb.
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Participants
  High | 4 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0
  Medium | 9 | 1 | 3 | 2 | 1 | 2 | 4 | 0 | 0 | 0
  Low | 13 | 3 | 12 | 20 | 12 | 6 | 22 | 11 | 13 | 8
  Unknown | 16 | 0 | 7 | 1 | 7 | 3 | 9 | 10 | 3 | 1

33. Secondary Outcome: Number of Participants With Different DNA Damage Repair (DDR) Status at Baseline
Description: DDR defect positive was determined by presence of one or more pathogenic or likely pathogenic mutations in tissue, DNA and/or blood samples.
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
Number analyzed (Participants) | 42 | 5 | 22 | 23 | 20 | 11 | 40 | 21 | 18 | 9
Participants
  Positive | 12 | 3 | 10 | 19 | 5 | 10 | 18 | 7 | 16 | 8
  Negative | 30 | 2 | 12 | 4 | 15 | 1 | 22 | 13 | 2 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From start of the treatment up to 90 days post last dose of study treatment (maximum of 5.2 years approximately), TEAEs and Serious TEAEs: from first dose of any study treatment and up to 30 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first (maximum of 5.2 years approximately).
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. Safety set was evaluated. The safety analysis set included all participants who received at least 1 dose of study drug. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD | Phase 2: Cohort A1 (NSCLC) | Phase 2: Cohort A2 (NSCLC DDR+) | Phase 2: Cohort B1 (TNBC) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) | Phase 2: Cohort C1 (OVC) | Phase 2: Cohort C2 (OVC BRCA-mutated) | Phase 2: Cohort D (UC) | Phase 2: Cohort E1 (mCRPC) | Phase 2: Cohort E2 (mCRPC DDR+) | Phase 2: Cohort F (BRCA/ATM-mutated)
All-Cause Mortality (participants affected / at risk) | 6/12 | 33/42 | 3/5 | 16/22 | 16/23 | 11/20 | 6/11 | 26/40 | 16/21 | 14/18 | 7/9
Serious Adverse Events (participants affected / at risk) | 1/12 | 16/42 | 2/5 | 7/22 | 5/23 | 9/20 | 2/11 | 16/40 | 5/21 | 9/18 | 4/9
Other Adverse Events (participants affected / at risk) | 12/12 | 41/42 | 5/5 | 21/22 | 22/23 | 20/20 | 10/11 | 38/40 | 21/21 | 16/18 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD (N=12) | Phase 2: Cohort A1 (NSCLC) (N=42) | Phase 2: Cohort A2 (NSCLC DDR+) (N=5) | Phase 2: Cohort B1 (TNBC) (N=22) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) (N=23) | Phase 2: Cohort C1 (OVC) (N=20) | Phase 2: Cohort C2 (OVC BRCA-mutated) (N=11) | Phase 2: Cohort D (UC) (N=40) | Phase 2: Cohort E1 (mCRPC) (N=21) | Phase 2: Cohort E2 (mCRPC DDR+) (N=18) | Phase 2: Cohort F (BRCA/ATM-mutated) (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3 | 2 | 0 | 0 | 3 | 0 | 0 | 1
Autoimmune neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 2
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Avelumab 800 mg Q2W + Talazoparib 1 mg QD (N=12) | Phase 2: Cohort A1 (NSCLC) (N=42) | Phase 2: Cohort A2 (NSCLC DDR+) (N=5) | Phase 2: Cohort B1 (TNBC) (N=22) | Phase 2: Cohort B2 (BC HR+ HER2- DDR+) (N=23) | Phase 2: Cohort C1 (OVC) (N=20) | Phase 2: Cohort C2 (OVC BRCA-mutated) (N=11) | Phase 2: Cohort D (UC) (N=40) | Phase 2: Cohort E1 (mCRPC) (N=21) | Phase 2: Cohort E2 (mCRPC DDR+) (N=18) | Phase 2: Cohort F (BRCA/ATM-mutated) (N=9)
Anaemia (Blood and lymphatic system disorders) | 8 | 28 | 4 | 18 | 10 | 12 | 7 | 31 | 15 | 10 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 7 | 0 | 3 | 1 | 4 | 0 | 5 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 4 | 0 | 5 | 0 | 4 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 10 | 2 | 6 | 4 | 4 | 2 | 6 | 3 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 15 | 1 | 9 | 2 | 9 | 4 | 16 | 6 | 3 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hypophosphatasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 1 | 0 | 3 | 2 | 1 | 1 | 1 | 0 | 0
Immune-mediated hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 8 | 0 | 2 | 2 | 4 | 0 | 4 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 5 | 7 | 0 | 0 | 4 | 4 | 2 | 4 | 3 | 2 | 2
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 17 | 4 | 8 | 10 | 11 | 8 | 14 | 10 | 5 | 6
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 5 | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 3 | 3 | 2 | 4
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 7 | 0 | 2 | 4 | 2 | 3 | 8 | 2 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 3 | 3 | 1 | 0 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 6 | 3 | 5 | 4 | 3 | 4 | 7 | 5 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 8 | 1 | 2 | 5 | 7 | 3 | 7 | 4 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 2 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 14 | 0 | 10 | 11 | 14 | 6 | 12 | 8 | 6 | 2
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue pigmentation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0 | 4 | 6 | 4 | 4 | 2 | 6 | 3 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 6 | 0 | 2 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 1 | 1 | 1 | 1 | 6 | 4 | 2 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 1 | 2 | 4 | 2 | 2 | 2 | 0 | 1
Amylase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 3 | 2 | 1 | 1 | 3 | 1 | 1 | 3 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 2 | 3 | 2 | 1 | 3 | 1 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 9 | 1 | 3 | 2 | 3 | 1 | 4 | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 1 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 4 | 0 | 7 | 4 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 4 | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 5 | 1 | 3 | 0 | 3 | 1 | 3 | 2 | 2 | 4
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 4 | 1 | 1 | 1 | 4 | 1 | 2 | 3 | 1 | 3
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 2 | 3 | 3 | 0 | 3 | 4 | 2 | 2
Neutrophil count decreased (Investigations) | 2 | 2 | 0 | 1 | 3 | 5 | 10 | 5 | 3 | 2 | 1
Platelet count decreased (Investigations) | 1 | 3 | 1 | 4 | 4 | 5 | 7 | 7 | 8 | 7 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 4 | 1 | 0 | 1 | 1 | 4 | 1 | 9 | 4 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 18 | 2 | 4 | 3 | 5 | 1 | 5 | 5 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1 | 0 | 4 | 0 | 4 | 2 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 5 | 2 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 2 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 4 | 1 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 4 | 2 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 2 | 6 | 2 | 2 | 8 | 2 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1 | 1 | 8 | 5 | 2 | 5 | 4 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 4 | 1 | 3 | 2 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 8 | 1 | 1 | 2 | 4 | 2 | 3 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 3 | 2 | 0 | 5 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 7 | 0 | 4 | 4 | 2 | 4 | 3 | 2 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 0 | 2 | 2 | 2 | 3 | 7 | 1 | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 17 | 1 | 9 | 2 | 7 | 3 | 8 | 2 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 3 | 3 | 3 | 3 | 1 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03330405/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03330405/SAP_001.pdf